CLINICAL TRIAL: NCT00180388
Title: Comparison of Clinical and Economical Parameters of Healing in Different Vein Harvesting Methods During Aortocoronary CABG
Brief Title: VENEK: Healing in Different Vein Harvesting Methods During Aortocoronary Coronary Artery Bypass Graft Surgery (CABG)
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: terminated for logistical reasons
Sponsor: Boston Scientific Corporation (Industry)
Collaborators: Herzzentrum Dresden (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Version vom 30.01.2004
Record Dates: First submitted 2005-09-12; First posted 2005-09-16 (Estimated); Last update posted 2016-09-01 (Estimated); Status verified 2007-03

CONDITIONS: Coronary Artery Disease
Keywords: cardiovascular system; veins; saphenous vein
MeSH Terms: conditions — Coronary Artery Disease

ARMS (2):
- Endoscopic vein harvesting (Experimental): Harvesting of vein for coronary artery bypass grafting using endoscopy to visualize the vein
  Interventions: Procedure: endoscopic vein harvesting
- Open Vein harvesting (Active Comparator): Harvesting of vein for coronary artery bypass grafting without endoscopy
  Interventions: Procedure: open vein harvesting

INTERVENTIONS:
Procedure: endoscopic vein harvesting
  Arms: Endoscopic vein harvesting
Procedure: open vein harvesting
  Arms: Open Vein harvesting

SUMMARY:
The VENEK trial is a randomized, prospective trial to compare economic parameters, quality of life and wound healing after endoscopic vein harvesting versus open vein harvesting.

DETAILED DESCRIPTION:
The VENEK trial is a randomized, prospective trial to compare economic parameters, quality of life and wound healing after endoscopic vein harvesting versus open vein harvesting.

ELIGIBILITY:
Inclusion Criteria:

* Age over 60 years
* Admission at Herzzentrum Dresden - Herzchirurgie for bypass-operation (OP) with planned veinectomy
* Eligibility for different modes of planned intervention according to study protocol
* Signed patient informed consent

Exclusion Criteria:

* Varicose crural veins
* Emergency patients
* Combined operational procedures
* Preoperative complete immobilization

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2004-05; Primary Completion 2006-06 (Actual); Study Completion 2006-06 (Actual)

PRIMARY OUTCOMES:
Evaluation of the economic differences between methods of treatment | up to 2 months
  Follow-up until wound healing

SECONDARY OUTCOMES:
Evaluation of the outcome in quality of life (questions according to the protocol) and rate of disorders in wound healing | up to 2 months
  Follow-up until wound healing

CONTACTS AND LOCATIONS:
Overall Officials: Matschke Knaut, MD, Principal Investigator — TU Dresden, Medizinische Fakultät Carl Gustav Carus, Klinik für Kardiochirurgie, D - 01062 Dresden, Germany
Locations (2):
- Germany (2):
  - Klinik Bad Gottleuba, Bad Gottleuba
  - TU Dresden, Medizinische Fakultät Carl Gustav Carus, Klinik für Kardiochirurgie, Dresden